CLINICAL TRIAL: NCT02403895
Title: A Phase 2a, Multi-centre, Single-arm Trial of the Combination of AZD2014 and Weekly Paclitaxel in Patients With Relapsed or Refractory Squamous Non-Small Cell Lung Cancer After At Least One Line of Prior Therapy
Brief Title: AZD2014 and Weekly Paclitaxel in Squamous NSCLC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D2274C00001
Record Dates: First submitted 2015-03-07; First posted 2015-03-31 (Estimated); Results first posted 2018-07-03 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Squamous Non Small Cell Lung Cancer
MeSH Terms: interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-label AZD2014 (Experimental): Open-label AZD2014 given twice daily 3 days on, 4 days off during weekly paclitaxel
  Interventions: Drug: Open-label AZD2014; Drug: paclitaxel

INTERVENTIONS:
Drug: Open-label AZD2014 — Dual TORC1/TORC2 inhibitor
Drug: paclitaxel — Taxane

SUMMARY:
Open--label, phase 2a, multi-centre, single-arm study to assess the efficacy and safety of AZD2014 and weekly paclitaxel in patients with squamous non-small cell lung cancer (NSCLC)

DETAILED DESCRIPTION:
This is an open-label, phase 2a, multi-centre, single-arm study to assess the efficacy and safety of the combination of AZD2014 and weekly paclitaxel in patients with squamous non-small cell lung cancer (NSCLC) that is relapsed or refractory to conventional treatment after at least 1 prior treatment with standard of care (SOC) and for whom weekly paclitaxel treatment is an appropriate treatment choice.

The study will simultaneously enrol patients to the following two groups. Group A (intensive PK) will enrol 10 evaluable patients for an intra-patient evaluation of the impact of paclitaxel on exposure to AZD2014, and the impact of AZD2014 on exposure to paclitaxel via intensive PK sampling and non-compartmental PK analysis techniques (NCA). Group B (sparse PK) will enrol 30 patients and sparse sampling and population PK modelling techniques will be employed to estimate exposure to AZD2014 when administered in combination with a weekly paclitaxel dosing regimen. The efficacy and safety of the AZD2014 and weekly paclitaxel combination will be evaluated in all 40 patients using RECIST 1.1, observation of AEs/SAEs and use of conventional safety parameters.

Eligible patients will receive study treatment consisting of a single weekly paclitaxel infusion (80 mg/m2) on Day 1 of each week and twice daily (BD) 50 mg doses of AZD2014 on the first 3 days each week for 6 weeks [except Group A patients in Week 1 of Cycle 1 who will take 50 mg BD doses of AZD2014 on Days 3, 4 and 5 (or Days 4, 5 and 6) to accommodate PK sampling], followed by a break from treatment when no paclitaxel or AZD2014 will be given. This 7-week schedule composes one cycle of treatment. AZD2014 will be administered as oral tablets to fasted patients (i.e., no food 2 hours before and 1 hour after each dose). Patients will receive up to 6 cycles of paclitaxel, although additional cycles of paclitaxel may be given if deemed appropriate by the Investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven squamous non-small cell lung cancer (NSCLC) where treatment with weekly paclitaxel is an appropriate treatment option.
2. Relapsed or refractory disease after at least one line of prior therapy. Subjects must have previously received appropriate line(s) of standard of care (SOC) treatment.
3. Measurable disease by RECIST v1.1 criteria
4. Life expectancy of at least 12 weeks.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Exclusion Criteria:

1. Radiotherapy (except for palliative reasons), chemotherapy, endocrine therapy, or immunotherapy during the previous 3 weeks (4 weeks for investigational medicinal products and 6 weeks for nitrosoureas and Mitomycin-C) before treatment.
2. Ongoing toxic manifestations of previous treatments. Exceptions to this are alopecia or Grade 1 toxicities which, in the opinion of the Investigator, should not exclude the patient.
3. Known leptomeningeal involvement, brain metastases or spinal cord compression.
4. History of hypersensitivity (> Grade 2) to active or inactive excipients of AZD2014, drugs containing Cremophor, taxanes or structurally/chemically similar drugs
5. Current refractory nausea and vomiting, chronic gastrointestinal disease, inability to swallow formulated product or previous significant bowel resection that would preclude adequate absorption of AZD2014
6. Patients with Diabetes Type I or uncontrolled Type II (HbA1c > 59 mmol/mol assessed locally) as judged by the Investigator
7. Major surgery within 4 weeks prior to entry to the study (excluding placement of vascular access), or minor surgery within 2 weeks of entry into the study and from which the patient has not yet recovered
8. Adequate hematologic function independent of transfusion and growth factor support for at least 7 days prior to screening (with the exception of pegylated G-CSF (pegfilgrastim) and darbepoetin which require at least 14 days prior to screening), defined as:

   * Absolute neutrophil count 1500 cells/mm3 (1.5 x 109/L)
   * Platelet count 100.000 cells/mm3 (100 x 109/L)
   * Haemoglobin 9.0 g/dL
9. Adequate hepatic and renal function defined as:

   * Serum aspartate transaminase (AST) or alanine transaminase (ALT) 2.5 x upper limit of normal (ULN) if no demonstrable liver metastases or 5 x ULN in the presence of liver metastases
   * Alkaline phosphatase (ALP) < 5 x ULN
   * Serum bilirubin 1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin)
   * Estimated Creatinine Clearance 50 ml/min (Cockcroft-Gault) or serum creatinine 1.5 x ULN

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-04-15 (Actual); Primary Completion 2016-12-29 (Actual); Study Completion 2016-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chandra P Belani, MD, Principal Investigator — Hershey Medical Center
Locations (7):
- United States (4):
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Hershey, Pennsylvania
  - Research Site, Dallas, Texas
- Research Site, Gauting, Germany
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Girona

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled: 15 April 2015 Last subject last visit: 29 December 2016 The study was performed at 7 centres: 4 USA, 2 Spain, 1 Germany Patient population: Patients with squamous non-small cell lung cancer with relapsed or refractory disease for whom weekly paclitaxel is an appropriate treatment choice
Pre-assignment Details: 11 patients were enrolled Patients were assigned to treatment if they met all of the inclusion criteria and none of the exclusion criteria.
Period: Overall Study
Arm/Group | Open-label AZD2014
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Open-label AZD2014
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Have a Partial Response or Complete Response Through Measurement of Tumour Lesion Sizes
Description: Calculation of the percentage of patient who have a Complete Response or Partial Response to treatment which is confirmed by a repeat assessment 4 weeks later
Time Frame: From first dose until disease progression (Approximately 3 months)
Population: Analysis Set: Evaluable for efficacy set. All dosed patients with a baseline tumour assessment
Measure: Number (90% Confidence Interval); unit: Percentage
Arm/Group | Open-label AZD2014
Number analyzed (Participants) | 11
Percentage
  Complete Response (CR) | 0 [0 to 23.8]
  Partial Response (PR) | 0 [0 to 23.8]

2. Secondary Outcome: Number of Patients Who Experienced at Least One Adverse Event (AE) or Serious Adverse Event (SAE)
Description: The safety and tolerability of AZD2014 with weekly paclitaxel as assessed with the collection of Adverse Events and Serious Adverse Events as reported during clinic visits. In addition, clinical assessments were made throughout the on treatment period including blood test for chemistry, haematology, and blood clotting. In addition to clinical observations such as vital signs, and cardiac function through the use of ECG.
  Any findings from the above assessments which were considered to be abnornal and clinically significant by the doctor were reported as (AEs or SAEs).
Time Frame: Informed consent until end of safety follow up (Approx 10 months if all treatment cycles are completed)
Measure: Number; unit: Count of Participants
Arm/Group | Open-label AZD2014
Number analyzed (Participants) | 11
Count of Participants
  Adverse Event (AE) | 11
  Serious Adverse Event (SAE) | 4

3. Secondary Outcome: Overall Survival: Median Number of Days Between the First Dose and End of Life Due to Any Cause
Description: Assessment of the duration of overall survival in weeks through direct patient follow-up. Any patient not known to have died at the time of analysis censored at the last recorded date the patient was known to be alive
Time Frame: From first dose until end of life (Approx 9 months)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Open-label AZD2014
Number analyzed (Participants) | 11
Days | 104 [27 to 164]

4. Secondary Outcome: Best Objective Response: Number of Patients Who Experienced a Best Response of Complete Response (CR), Partial Response (PR), Stable Disease (SD), Progressive Disease (PD), Not-Evaluable (NE), Through Measurement of Tumour Lesion Sizes.
Description: Per Response Evaluation Criteria In Solid Tumours (RECIST v1.1) for target lesions assessed through imaging (CT or MRI scan) or clinical examination; Complete Response (CR): Disappearance of all target lesions; Partial Response (PR) >=30% decrease in sum of target lesion longest diameter; Progressive Disease >=20% increase in sum of target lesion longest diameter; Stable Disease (SD) increase or decrease amounting to neither PR or PD. Overall tumour assessment based on quantitative assessment of target lesions and qualitative assessment of non-target lesions in line with RECIST criteria.
Time Frame: From Baseline until Disease Progression (Approx 3 months)
Measure: Number; unit: Count of Participants
Arm/Group | Open-label AZD2014
Number analyzed (Participants) | 11
Count of Participants
  PD | 6
  SD | 5
  PR | 0
  CR | 0

5. Secondary Outcome: Duration of Response: Median Number of Days From the Date of First Documented Response Until the Date of Documented Progression Through Measurement of Tumour Lesion Sizes
Description: Assessment of the duration of tumour response through assessment of tumour lesions by RECIST 1.1 criteria. Response is defined as the point at which the criteria for Partial Response (PR) was met) >=30% decrease in sum of target lesion longest diameter. Progression is defined as the point at which the criteria for Progressive Disease (PD) was met >=20% increase in sum of target lesion longest diameter, or until end of life.
Time Frame: From date of first documented response until documented progression or end of life in the absence of progression (Approx 3 months)
Population: No participant responded therefore no duration of response data to report
Arm/Group | Open-label AZD2014
Number analyzed (Participants) | 0

6. Secondary Outcome: Disease Control Rate: Percentage of Patients Who Achieve Partial Response, Complete Response or Stable Disease Through Assessment of Tumour Lesion Sizes
Description: Assessment of the disease control rate, percentage of patients who experience a response through assessment of tumour lesions by RECIST 1.1 criteria
Time Frame: From first dose until documented progression and at least 6 weeks after the start of treatment for assessment of Stable Disease - Assessed at 6, 13 and 20 Weeks
Measure: Number (80% Confidence Interval); unit: Percentage of patients
Arm/Group | Open-label AZD2014
Number analyzed (Participants) | 11
Percentage of patients
  Disease Control Rate at 6 Weeks | 45.5 [24.1 to 68.2]
  Disease Control Rate at 13 Weeks | 18.2 [4.9 to 41.5]
  Disease Control Rate at 20 Weeks | 18.2 [4.9 to 41.5]

7. Secondary Outcome: Change in Tumour Size: Median Percentage Change in Tumour Size in mm by Measurement of Tumour Lesion Sizes
Description: Assessment of the degree of tumour response through measurement of the change in tumour lesion sizes
Time Frame: From baseline until documented progression (Approx 3 months)
Measure: Median (Full Range); unit: % change
Arm/Group | Open-label AZD2014
Number analyzed (Participants) | 11
% change | 0.0 [-33.3 to 41.8]

8. Secondary Outcome: Progression Free Survival: Median Number of Days Between Start of Dosing Until Objective Disease Progression Through Measurement of Tumour Lesion Sizes
Description: Assessment of the duration of progression free survival through assessment of tumour lesions by RECIST 1.1 criteria
Time Frame: From date of first dose until documented progression or end of life (Approx 3 months)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Open-label AZD2014
Number analyzed (Participants) | 11
Days | 91 [15 to 98]

9. Secondary Outcome: Evaluate the Effect of the Combination of AZD2014 and Paclitaxel on Pharmacokinetics Assessment of Cmax
Description: To determine the effect of co-administration of paclitaxel on the PK of oral AZD2014 and the effect of co administration of oral AZD2014 on the PK of paclitaxel (Group A) by: PK parameters for each in the presence and absence of the other by intensive PK sampling and NCA techniques.
Time Frame: Assessment at multiple timepoints in Group A patients. Samples will be taken at pre-dose and at 10 further timepoints on day 1 and at pre-dose and 9 further timepoints on days 3 and 8
Population: Data insufficient for full PK parameter evaluation or comparisons made between AZD2014 and paclitaxel
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Open-label AZD2014
Number analyzed (Participants) | 2
ng/mL
  Paclitaxel Cmax | 2240 [1500 to 2980]
  AZD2014 Cmax | 1021 [741 to 1300]

10. Secondary Outcome: Estimated Pharmacokinetic Exposure to AZD2014 Through the Use of Population PK Modelling
Description: Group B patients: PK parameters for AZD2014 estimated from a sparse PK sampling regimen and use of population PK modelling techniques (may be reported outside the clinical study report (CSR))
Time Frame: Assessment at multiple timepoints in Group B patients between study day 1 and day 3. Samples will be taken at 3 points on day 1 and at predose and at a further 2 points on day 3
Population: The exposure of AZD2014 could not be estimated using a population PK model because there were insufficient subjects with intensive PK sampling (n=2) to develop at population PK model
Arm/Group | Open-label AZD2014
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the time of informed consent throughout the treatment period until the end of the follow-up period. The follow-up period if defined as 28 days after study treatment is discontinued for a given patient. Total duration of collection period = approximately 10 months if all cycles and follow-up period is completed.
Description: Adverse events were assessed systematically through clinical review, and collection of laboratory assessment, physical examination, performance status, ECHO/MUGA and ECG. Patients attended the clinic for assessment on a weekly basis
Arm/Group | Open-label AZD2014
All-Cause Mortality (participants affected / at risk) | 9/11
Serious Adverse Events (participants affected / at risk) | 4/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label AZD2014 (N=11)
Cellulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Seizure (Nervous system disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label AZD2014 (N=11)
Pneumonia (Infections and infestations) | 1
Anaemia (Blood and lymphatic system disorders) | 3
Neuropathy Peripheral (Nervous system disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 2
Fatigue (General disorders) | 4
Fungal Infection (Infections and infestations) | 1
Lower Respiratory Tract Infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Increased appetite (Metabolism and nutrition disorders) | 1
Depression (Psychiatric disorders) | 1
Eating disorder symptom (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Headache (Nervous system disorders) | 1
Nerve compression (Nervous system disorders) | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Papule (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Mucosal Inflammation (General disorders) | 1
Weight decreased (Investigations) | 1
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1

LIMITATIONS AND CAVEATS:
Sponsor and Investigator decision was taken to terminate further recruitment into the study due to lack of observed responses rendering it futile to continue. As such, an abbreviated Clinical Study Report was produced based on data from 11 patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other